CLINICAL TRIAL: NCT04797507
Title: SHR-1210, a Novel Anti-PD-1 Antibody, in Combination With Anlotinib As Second-line or Above Treatment in Patients With Advanced or Metastatic Esophageal Squamous Cell Cancer: a Phase II Study
Brief Title: SHR-1210 in Combination With Anlotinib in Patients With Advanced or Metastatic Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2681
Record Dates: First submitted 2021-02-25; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: SHR-1210; Anlotinib; Advanced Esophageal Squamous Cell Cancer
MeSH Terms: interventions — camrelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): SHR-1210 plus Anlotinib
  Interventions: Drug: SHR-1210 plus Anlotinib

INTERVENTIONS:
Drug: SHR-1210 plus Anlotinib — SHR-1210: a novel anti-PD-1 antibody Anlotinib: a multi-kinase inhibitor

SUMMARY:
This study was designed to explore the clinical efficacy of SHR-1210 in combined with Anlotinib in the treatment of second- or above- line advanced or metastatic esophageal squamous cell cancer patients, in order to find a better therapy strategy for esophageal squamous cell cancer patients.

DETAILED DESCRIPTION:
This is a prospective, phase II, single-arm clinical trial. Advanced or metastatic esophageal squamous cell cancer(ESCC) patients progressed after 1st systematic treatment are treated with SHR-1210 and Anlotinib. SHR-1210 was given intravenously(200mg d1 Q2w), combined with Anlotinib orally, 12 mg d1-14 Q3w. The hypothesis: The objective response rate in SHR-1210 combined with Anlotinib can reach 40% as second-line or above treatment of advanced or metastatic ESCC patients. The primary endpoint is objective response rate (ORR) and the secondary endpoint is disease control rate (DCR), overall survival (OS), progression-free survival (PFS), and safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 years to 75 years, male or female.
2. Histologically or cytologically confirmed squamous cell carcinoma of the esophagus, locally advanced, unresectable, recurrent or metastatic disease.
3. Progressed after first-line chemotherapy.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
5. Newly acquired or archived tumor tissue samples can be obtained.
6. Eastern Collaborative Oncology Group (ECOG) Performance Status ≤ 1
7. Life expectancy >12 weeks.
8. Adequate organ function.
9. For females of child bearing potential, a negative urine or serum pregnancy test result within 1 week before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study until 4 months after the last dose of any of the drugs in the study.
10. Willing and able to follow the study protocol and follow-up procedures for treatment and follow-up.
11. Willing and able to provide written informed consent.

Exclusion Criteria:

Patients should not be selected for this clinical study if they have any of the following conditions:

1. Abnormal coagulation function , with bleeding tendency or receiving thrombolytic or anticoagulant therapy. Note: Low-dose heparin (60,000-12,000 U/day for adults) or low-dose aspirin (≤100mg/day) are permitted for prophylactic purposes if INR≤1.5.
2. The arterial/venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis, pulmonary embolism, etc, occurred within 6 months before administration.
3. Clinically significant hemoptysis occurred within 3 months before medication (hemoptysis > 50ml per day); Or clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, baseline fecal occult blood ++ or above, or vasculitis, etc.
4. Subjects with any active, known or suspected autoimmune disease or history of autoimmune disease.
5. Received systemic steroid therapy within 3 days of the first dose of study medication.
6. Received a live vaccine within 4 weeks of the first dose of study medication.
7. Major surgery received or severe traumatic injury, fracture, or ulcer occurred within 4 weeks of the first dose of study medication.
8. Imaging (CT or MRI) showed that the distance of the tumor lesion from great vessels was less than 5 mm, or invasion of local great vessels, or central tumor with high blood risk; Or there is obvious lung cavity or necrotizing tumor. Uncontrolled clinically significant systemic diseases, including active infection, unstable angina, angina occurred within 3 months,≥ NYHA II congestive heart failure, myocardial infarction occurred within 6 months, severe arrhythmia, liver, kidney, or metabolic disease.
9. Pregnant or lactating female.
10. Participate in other clinical trials currently or within 4 weeks prior to enrollment.
11. Receiving other anti-cancer drugs (including anti-cancer traditional chinese medicine).
12. Familial, sociological or geographical conditions that, in the clinical judgment of the Principal Investigator, do not permit compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
ORR based on RECIST v1.1 | 12 months
  Objective response rate based on RECIST v1.1 by investigators

SECONDARY OUTCOMES:
DCR based on RECIST v1.1 | 12 months
  Disease control rate based on RECIST v1.1 by investigators
Overall survival | 24 months
  Overall survival based on RECIST v1.1 by investigators
Progression free survival | 12 months
  Progression free survival based on RECIST v1.1 by investigators
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  Safety and tolerance by investigators

IPD SHARING:
Plan to Share IPD: No